CLINICAL TRIAL: NCT06419127
Title: Embryo Assessment Utilizing Timelapse Imaging in Conjunction With Preimplantation Genetic Testing for Aneuploidy With Next Generation Sequencing
Status: Enrolling by invitation | Type: Observational
Sponsor: Gattaca Genomics (Industry)
Responsible Party: Sponsor
Other Study IDs: GG1001
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Infertility, Female; Infertility, Male; Infertility; IVF; Aneuploidy
Keywords: ivf; infertility; pgt; embryo
MeSH Terms: conditions — Infertility, Female; Infertility, Male; Infertility; Aneuploidy; Long Qt Syndrome 3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The piece of the embryo that is utilized for PGT will be amplified, analyzed, and maintained according to standard operating procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile patients: Infertile patients undergoing IVF with PGT.
  Interventions: Diagnostic Test: Timelapse incubation and PGT

INTERVENTIONS:
Diagnostic Test: Timelapse incubation and PGT — Patients will have their embryos cultured in a timelapse incubator and their PGT results will be compared to the data collected during timelapse incubation.

SUMMARY:
The goal of this observational study is to discern if there is a relationship between timelapse imagery of human oocytes/embryos and PGT results.

Embryos of patients that are undergoing PGT will be placed into a timelapse incubator. The data obtained by the timelapse incubator will be used in conjunction with the PGT data to determine any relationships.

DETAILED DESCRIPTION:
Timelapse imagery (TLI) is a multifaceted technology being utilized within the in vitro fertilization (IVF) space. With this technology it is possible to have a live, continuous video of embryo development from fertilization to implantation. During this live evaluation multiple datapoints can be extrapolated and used to determine embryo viability. Another technology used in the IVF space is preimplantation genetic testing for aneuploidy (PGT-A). With this technology, individual cells from the embryo are removed, amplified, and the chromosomal content of the cells is analyzed by next generation sequencing (NGS)-based technology, allowing the chromosomal content of the embryos to be determined prior to embryo transfer.

To date, no one has combined the data from both tools to try to advance the IVF field.

Gattaca Genomics is proposing utilizing the data obtained from TLI, in conjunction with the data obtained from PGT-A, to create a computer model that can accurately predict which embryos will lead to a successful outcome during IVF.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing IVF with PGT

Exclusion Criteria:

* patients undergoing IVF and not electing for PGT

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: All infertile patients undergoing IVF with PGT
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Time to first cleavage | 24 hours
  time of embryo to undergo first cleavage
Time to blastulation | 5-7 days
  time of embryo to form a blastocoel
Fertilization morphology | 24 hours
  the morphological appearance of the pronuclei
Embryo morphology | 2-7 days
  the morphological appearance of the embryos
Patient age | 0 days
  Patient age
Partner age | 0 days
  Partner age
Partner diagnosis | 0 days
  Partner diagnosis
Metabolomics of culture media | 7 days
  measurement of the spent culture media for amino acids, enzymes, and metabolites
AMH | 0 days
  antimullerian hormone level in female's blood
Days of stimulation | 0-15 days
  the number of days the patient underwent stimulation for IVF
Dosage of stimulation meds | 0-15 days
  the amount of stimulation meds the patient took during IVF treatment
Pregnancy | 2 weeks after transfer
  initial bhCG levels
Patient diagnosis | 0 days
  Number of patients with each specific diagnosis, including low ovarian reserve, PCOS, primary infertility, secondary infertility, endometrosis, and unknown infertility.
implantation | 4 weeks post transfer
  Number of patients that develope a sac within the uterus post transfer
fetal cardiac heartbeat | 6 weeks
  Number of patients that develop a fetal cardiac heartbeat after transfer
livebirth | approximately 9 months after transfer
  Number of patients that have a livebirth of an infant after IVF

CONTACTS AND LOCATIONS:
Locations (1):
- Gattaca Genomics, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with other researchers